CLINICAL TRIAL: NCT00071591
Title: Functional Skills Training for Late Life Schizophrenia
Brief Title: Rehabilitative Training for Older People With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Thomas L. Patterson, Professor, University of California, San Diego
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: R01MH062554 (NIH); R01MH062554 (NIH); DATR A4-GPS
Record Dates: First submitted 2003-10-29; First posted 2003-10-30 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Behavioral: Functional Adaptation Skills Training (FAST)

SUMMARY:
This study will evaluate the effectiveness of a rehabilitation program called Functional Adaptation Skills Training (FAST) in treating older patients with schizophrenia.

DETAILED DESCRIPTION:
People with schizophrenia often have problems functioning in everyday life. As people with schizophrenia get older, resources for effective health care and social services may become more limited. There is a need to develop effective rehabilitation programs that are sensitive to the special needs of older persons with schizophrenia.

Patients are randomly assigned to either 1 of 2 groups. The FAST group will involve 24 sessions of group intervention designed to enhance daily functioning of older patients with schizophrenia. The placebo group will involve participation in a psychosocial support group for an equivalent amount of time. Treatment is followed by 6 monthly maintenance sessions. Patients will be assessed at 6, 12, and 18 months after the study start. Assessments include clinical and functional measures.

ELIGIBILITY:
Inclusion Criteria:

* Have schizophrenia or schizoaffective disorder

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2001-07; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States